CLINICAL TRIAL: NCT03615417
Title: Effectiveness of High-Flow Nasal Cannula (HFNC) Preoxygenation in Obese Patients Undergoing General Anesthesia: A Randomised Controlled Trial
Brief Title: High-Flow Nasal Cannula (HFNC) Preoxygenation in Obese Patients Undergoing General Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasme University Hospital (Other)
Responsible Party: Principal Investigator, Francesco Ricottilli, MD, Resident, Department of Anesthesiology, Erasme University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SRB-201712-161; B406201834736 (Other: CCB - Comité consultatif de Bioéthique de Belgique); P2018/067 (Other: Erasme - ULB Ethics Committee)
Record Dates: First submitted 2018-07-30; First posted 2018-08-03 (Actual); Last update posted 2018-11-19 (Actual); Status verified 2018-11

CONDITIONS: Preoxygenation; Anesthesia; Obesity
MeSH Terms: conditions — Obesity | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HFNC - High Flow Nasal Cannula (Experimental): Participants are preoxygenated by High Flow Nasal Cannula (HFNC) OptiFlow.
  Interventions: Device: High Flow Nasal Cannula (HFNC)
- FM - FaceMask (Active Comparator): Participants are preoxygenated by standard anesthesia FaceMask.
  Interventions: Device: Standard anesthesia FaceMask (FM)

INTERVENTIONS:
Device: High Flow Nasal Cannula (HFNC) — Preoxygenation trough High Flow Nasal Cannula (HFNC) at 100% FiO2, 50 liters/min and closed mouth.
  After Rapid Sequence Induction (RSI), maintenance of apnea with HFNC at 100% FiO2, 70 liters/min and jaw thrust.
  At time of peripheral oxygen saturations (SpO2) decreases by 2% or after 10 minutes of apnea, the participant is intubated.
  Other Names: THRIVE; OptiFlow
  Arms: HFNC - High Flow Nasal Cannula
Device: Standard anesthesia FaceMask (FM) — Preoxygenation trough standard anesthesia FaceMask (FM) at 100% FiO2, 12 liters/min, CPAP 7 cmH2O.
  After Rapid Sequence Induction (RSI), maintenance of apnea without mask. At time of peripheral oxygen saturations (SpO2) decreases by 2% or after 10 minutes of apnea, the participant is intubated.
  Arms: FM - FaceMask

SUMMARY:
This study aims to evaluate the effectiveness of the High Flow Nasal Cannula (HFNC) for the preoxygenation of obese patients undergoing a general anesthesia. The HFNC interface is compared to a standard anesthesia FaceMask (FM) preoxygenation with Continuous Positive Airway Pressure (CPAP), the current gold standard procedure for obese induction.

The interest of HFNC preoxygenation is to increase the "safe apnea time" before critical arterial desaturation, useful in the management of difficult airways, especially in subjects with reduced respiratory reserves such as the obese.

ELIGIBILITY:
Inclusion Criteria:

* Surgery with the need for general anesthesia with muscle relaxation
* ASA (American Society of Anesthesiologists) physical status score II-III
* BMI > 35

Exclusion Criteria:

* Severe respiratory disease (acute respiratory failure, Chronic obstructive pulmonary disease COPD, parenchymal pneumopathies,...)
* Severe nasal pathology (malformation, stenosis)
* Criteria or previous difficult intubation
* BMI > 50
* Chest circumference > 150cm
* Implanted electronic device (pacemaker, neurostimulator, ...)
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-04-19 (Actual); Primary Completion 2018-09-07 (Actual); Study Completion 2018-09-07 (Actual)

PRIMARY OUTCOMES:
Functional Residual Capacity (FRC) variation | 20 minutes
  The difference of FRC, estimated by lung Electrical Impedance Tomography (EIT), during general anesthesia induction (from a base period to the mechanical ventilation).

SECONDARY OUTCOMES:
Time of safe apnea | 20 minutes
  The time (seconds) of apnea following preoxygenation and muscle relaxation before to peripheral oxygen saturations (SpO2) decreases by 2%, or the apnea time reaches 600 seconds.
Lowest SpO2 | 20 minutes
  The lowest SpO2 (%) during general anesthesia induction (from a base period to the mechanical ventilation).
Preoxygenation Comfort | 6 hours
  The subjective comfort of the patient during the preoxygenation, expressed with a 0-5 scale at Post Anesthesia Care Unit (PACU) discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Ricottilli, MD, Principal Investigator — Erasme University Hospital
Locations (1):
- Erasme University Hospital, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Drake MG. High-Flow Nasal Cannula Oxygen in Adults: An Evidence-based Assessment. Ann Am Thorac Soc. 2018 Feb;15(2):145-155. doi: 10.1513/AnnalsATS.201707-548FR. PMID 29144160
- [Background] Okuda M, Tanaka N, Naito K, Kumada T, Fukuda K, Kato Y, Kido Y, Okuda Y, Nohara R. Evaluation by various methods of the physiological mechanism of a high-flow nasal cannula (HFNC) in healthy volunteers. BMJ Open Respir Res. 2017 Jul 20;4(1):e000200. doi: 10.1136/bmjresp-2017-000200. eCollection 2017. PMID 29071075
- [Background] Ang KS, Green A, Ramaswamy KK, Frerk C. Preoxygenation using the Optiflow system. Br J Anaesth. 2017 Mar 1;118(3):463-464. doi: 10.1093/bja/aex016. No abstract available. PMID 28203758
- [Background] White LD, Melhuish TM, White LK, Wallace LA. Apnoeic oxygenation during intubation: a systematic review and meta-analysis. Anaesth Intensive Care. 2017 Jan;45(1):21-27. doi: 10.1177/0310057X1704500104. PMID 28072931
- [Background] Mir F, Patel A, Iqbal R, Cecconi M, Nouraei SA. A randomised controlled trial comparing transnasal humidified rapid insufflation ventilatory exchange (THRIVE) pre-oxygenation with facemask pre-oxygenation in patients undergoing rapid sequence induction of anaesthesia. Anaesthesia. 2017 Apr;72(4):439-443. doi: 10.1111/anae.13799. Epub 2016 Dec 30. PMID 28035669
- [Background] Bauchmuller KB, Glossop AJ, De Jong A, Jaber S. Combining high-flow nasal cannula oxygen and non-invasive ventilation for pre-oxygenation in the critically ill: is a double-pronged approach warranted? : Discussion on article "Apnoeic oxygenation via high-flow nasal cannula oxygen combined with non-invasive ventilation preoxygenation for intubation in hypoxaemic patients in the intensive care unit: the single-centre, blinded, randomised controlled OPTINIV trial". Intensive Care Med. 2017 Feb;43(2):288-290. doi: 10.1007/s00134-016-4635-6. Epub 2016 Dec 8. No abstract available. PMID 27933345
- [Background] Jaber S, Monnin M, Girard M, Conseil M, Cisse M, Carr J, Mahul M, Delay JM, Belafia F, Chanques G, Molinari N, De Jong A. Apnoeic oxygenation via high-flow nasal cannula oxygen combined with non-invasive ventilation preoxygenation for intubation in hypoxaemic patients in the intensive care unit: the single-centre, blinded, randomised controlled OPTINIV trial. Intensive Care Med. 2016 Dec;42(12):1877-1887. doi: 10.1007/s00134-016-4588-9. Epub 2016 Oct 11. PMID 27730283
- [Background] Doyle AJ, Stolady D, Mariyaselvam M, Wijewardena G, Gent E, Blunt M, Young P. Preoxygenation and apneic oxygenation using Transnasal Humidified Rapid-Insufflation Ventilatory Exchange for emergency intubation. J Crit Care. 2016 Dec;36:8-12. doi: 10.1016/j.jcrc.2016.06.011. Epub 2016 Jun 23. PMID 27546740
- [Background] Ward JJ. High-flow oxygen administration by nasal cannula for adult and perinatal patients. Respir Care. 2013 Jan;58(1):98-122. doi: 10.4187/respcare.01941. PMID 23271822
- [Background] Corley A, Caruana LR, Barnett AG, Tronstad O, Fraser JF. Oxygen delivery through high-flow nasal cannulae increase end-expiratory lung volume and reduce respiratory rate in post-cardiac surgical patients. Br J Anaesth. 2011 Dec;107(6):998-1004. doi: 10.1093/bja/aer265. Epub 2011 Sep 9. PMID 21908497
- [Background] Parke R, McGuinness S, Eccleston M. Nasal high-flow therapy delivers low level positive airway pressure. Br J Anaesth. 2009 Dec;103(6):886-90. doi: 10.1093/bja/aep280. Epub 2009 Oct 20. PMID 19846404
- [Background] Kostic P, LoMauro A, Larsson A, Hedenstierna G, Frykholm P, Aliverti A. Specific anesthesia-induced lung volume changes from induction to emergence: a pilot study. Acta Anaesthesiol Scand. 2018 Mar;62(3):282-292. doi: 10.1111/aas.13026. Epub 2017 Nov 3. PMID 29105056
- [Background] Nimmagadda U, Salem MR, Crystal GJ. Preoxygenation: Physiologic Basis, Benefits, and Potential Risks. Anesth Analg. 2017 Feb;124(2):507-517. doi: 10.1213/ANE.0000000000001589. PMID 28099321
- [Background] Fraser JF, Spooner AJ, Dunster KR, Anstey CM, Corley A. Nasal high flow oxygen therapy in patients with COPD reduces respiratory rate and tissue carbon dioxide while increasing tidal and end-expiratory lung volumes: a randomised crossover trial. Thorax. 2016 Aug;71(8):759-61. doi: 10.1136/thoraxjnl-2015-207962. Epub 2016 Mar 25. PMID 27015801
- [Background] Harbut P, Gozdzik W, Stjernfalt E, Marsk R, Hesselvik JF. Continuous positive airway pressure/pressure support pre-oxygenation of morbidly obese patients. Acta Anaesthesiol Scand. 2014 Jul;58(6):675-80. doi: 10.1111/aas.12317. Epub 2014 Apr 16. PMID 24738713
- [Background] Nakahashi S, Gando S, Ishikawa T, Wada T, Yanagida Y, Kubota N, Uegaki S, Hayakawa M, Sawamura A. Effectiveness of end-expiratory lung volume measurements during the lung recruitment maneuver for patients with atelectasis. J Crit Care. 2013 Aug;28(4):534.e1-5. doi: 10.1016/j.jcrc.2012.11.003. Epub 2013 Jan 18. PMID 23337480
- [Background] Delay JM, Sebbane M, Jung B, Nocca D, Verzilli D, Pouzeratte Y, Kamel ME, Fabre JM, Eledjam JJ, Jaber S. The effectiveness of noninvasive positive pressure ventilation to enhance preoxygenation in morbidly obese patients: a randomized controlled study. Anesth Analg. 2008 Nov;107(5):1707-13. doi: 10.1213/ane.0b013e318183909b. PMID 18931236
- [Background] Baillard C, Fosse JP, Sebbane M, Chanques G, Vincent F, Courouble P, Cohen Y, Eledjam JJ, Adnet F, Jaber S. Noninvasive ventilation improves preoxygenation before intubation of hypoxic patients. Am J Respir Crit Care Med. 2006 Jul 15;174(2):171-7. doi: 10.1164/rccm.200509-1507OC. Epub 2006 Apr 20. PMID 16627862
- [Background] van Genderingen HR, van Vught AJ, Jansen JR. Estimation of regional lung volume changes by electrical impedance pressures tomography during a pressure-volume maneuver. Intensive Care Med. 2003 Feb;29(2):233-40. doi: 10.1007/s00134-002-1586-x. Epub 2002 Dec 14. PMID 12594585
- [Background] Hinz J, Hahn G, Neumann P, Sydow M, Mohrenweiser P, Hellige G, Burchardi H. End-expiratory lung impedance change enables bedside monitoring of end-expiratory lung volume change. Intensive Care Med. 2003 Jan;29(1):37-43. doi: 10.1007/s00134-002-1555-4. Epub 2002 Nov 20. PMID 12528020